CLINICAL TRIAL: NCT03107013
Title: An Open Label, Single-Dose, Single-Period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-BTD-001 in Healthy Male Subjects
Brief Title: A Study to Investigate the Mass Balance of BTD-001
Acronym: HV103
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Balance Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BTD-001 HV103
Record Dates: First submitted 2017-03-27; First posted 2017-04-11 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Molecular Mechanisms of Pharmacological Action
Keywords: Mass Balance; Phase 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-BTD-001 (Experimental)
  Interventions: Drug: [14C]-BTD-001

INTERVENTIONS:
Drug: [14C]-BTD-001 — Carbon-14 labeled BTD-001

SUMMARY:
This is a single-centre, open-label, non-randomised, single oral dose study in healthy male subjects to assess the mass balance recovery of carbon-14 (14C)-BTD-001.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged 30-65 years old
* BMI between18.0-35.0 kg/m2 unless investigator deems not clinically significant
* Regular daily bowel movements
* Provide written consent
* Agrees to protocol specified contraception

Exclusion Criteria:

* Received any investigational treatment within last 3 months
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week
* Current smokers and those who have smoked, including nicotine replacement or e-cigarates within the last 12 months.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
* Clinically significant abnormal lab results
* Positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Evidence of renal impairment at screening
* History of or current seizure disorder or history of syncope, unexplained loss of consciousness or seizure in the past 3 years
* Clinically significant medical/psychiatric history findings, or physical/neurological examination findings or significant history of or current suicidal ideation or behaviour
* History of or current significant pulmonary, cardiac, renal, hepatic, chronic respiratory, gastrointestinal, neurological or psychiatric disease, substance dependence, porphyria, malignancy (with exception of local cutaneous squamous or basal cell carcinomas or local cervical squamous cell cancer resolved after resection) or hypothyroidism
* Subjects with QT interval corrected for heart rate according to Fridericia's formula >450 msec
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than up to 4 g per day paracetamol) or herbal remedies
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery after a single dose of carbon-14 (14C)-BTD-001 | Maximum 12 days
  The percentage of radioactive dose of [14C] radiolabelled BTD-001 recovered in urine, faeces, and plasma
Metabolite Profiling | Maximum 12 days
  To provide plasma, urine and faecal samples for metabolite profiling and structural identification

SECONDARY OUTCOMES:
Determination of routes and rates of elimination of [14C]-BTD-001 | Maximum 12 days
  [14C]-BTD-001 metabolite profiling and structural identification in plasma, urine and faeces
Determination of the chemical structure of the "major" metabolites of [14C]-BTD-001 | Maximum 12 days
  Identification of the chemical structure of each metabolite accounting for more than 10% (by AUC) of circulating total radioactivity
Evaluation of whole blood:plasma concentration ratios for total radioactivity | Maximum 12 days
  To evaluate the extent of distribution of total radioactivity into blood cells
physical examination | Maximum 12 days
  Safety and tolerability of BTD-001 by assessing physical examination
safety laboratory tests | Maximum 12 days
  Safety and tolerability of BTD-001 by assessingsafety laboratory tests and AEs
Vital signs | Maximum 12 days
  Safety and tolerability of BTD-001 by assessing vital signs
ECGs | Maximum 12 days
  Safety and tolerability of BTD-001 by assessing ECGs
AEs | Maximum 12 days
  Safety and tolerability of BTD-001 by assessing physical examination AEs

OTHER OUTCOMES:
Cmax | Maximum 12 days
  Maximum Observed Plasma Concentration
tmax | Maximum 12 days
  time to reach maximum concentration
t1/2 | Maximum 12 days
  elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Nand Signh, MD, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided